CLINICAL TRIAL: NCT05434403
Title: Transauricular Vagus Nerve Stimulation in the Treatment of Chemotherapy-induced Peripheral Neuropathy: A Randomized Controlled Study
Brief Title: Transauricular Vagus Nerve Stimulation in the Treatment of Chemotherapy-induced Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, director of department of Anesthesiology and Pain medicine, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022PHB107-001
Record Dates: First submitted 2022-06-08; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: CIPN; Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham stimulation group (Placebo Comparator)
  Interventions: Device: sham vagus nerve stimulation
- stimulation group (Experimental)
  Interventions: Device: Vagus nerve stimulation

INTERVENTIONS:
Device: Vagus nerve stimulation — vagus nerve electrical stimulation through ear skin
  Arms: stimulation group
Device: sham vagus nerve stimulation — sham vagus nerve electrical stimulation through ear skin
  Arms: Sham stimulation group

SUMMARY:
Chemotherapy induced peripheral neuropathy is common in tumor patients receiving chemotherapy. Nowaday, CIPN is mainly treated with drugs, but the therapeutic effect is not satisfactory. Previous studies have found that inflammatory immune mechanism plays an important role in neuropathic pain. Vagus nerve stimulation can not only relieve pain by regulating the autonomic nervous system, but also participate in the immune response. Investigators hope that the treatment by vagus nerve electrical stimulation through ear skin can improve the pain and neurotoxicity scores of CIPN patient.If it is proved that vagus nerve stimulation can effectively treat CIPN, it will become a simple and safe non-drug treatment which has good application prospects.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is currently receiving chemotherapy drugs with neurotoxicity
2. New or worsening numbness and / or pain in the hands and / or feet, and no other cause explains the above symptoms

Exclusion Criteria:

1. Patients with sinus bradycardia, long QT syndrome, sick sinus syndrome or other arrhythmias, mental diseases, cardiac pacemakers or other electrical stimulation devices after implantation.
2. Patients taking analgesics due to pain in other parts of the body.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
NRS(numerical rating scale) | Day0
  0-10，0 =no pain, 10 = the most severe pain.
NRS(numerical rating scale) | Day3
  0-10，0 =no pain, 10 = the most severe pain.
NRS(numerical rating scale) | Day5
  0-10，0 =no pain, 10 = the most severe pain.
NRS(numerical rating scale) | Day8
  0-10，0 =no pain, 10 = the most severe pain.
NRS(numerical rating scale) | Day14
  0-10，0 =no pain, 10 = the most severe pain.
NRS(numerical rating scale) | Day30
  0-10，0 =no pain, 10 = the most severe pain.
NRS(numerical rating scale) | Day60
  0-10，0 =no pain, 10 = the most severe pain.
NRS(numerical rating scale) | Day90
  0-10，0 =no pain, 10 = the most severe pain.

SECONDARY OUTCOMES:
NCI-CTC v4.0 neurotoxicity classification | Day1,Day3,Day5,Day8,Day14,Day30,Day60,Day90
  Assess the degree of motor neurotoxicity and sensory neurotoxicity
QST( Quantitative Sensory Testing) | Day1,Day14
  left finger, thermal thretshold,thermal pain threshold,cold threshold,cold pain threshold,
IL-2，IL-4，IL-6，IL-10，IFN-γ，TNF-α | Day1,Day14
  Hematological examination to test the concentration of IL-2，IL-4，IL-6，IL-10，IFN-γ，TNF-α
Athens insomnia scale | Day1,Day8,Day14,Day30,Day60,Day90
  <4 No sleep disorder,4-6=Suspicious insomnia,>6=Insomnia
SF-12，Short From health survey -12 | Day1,Day8,Day14,Day30,Day60,Day90
  Calculate the Physical Component Summary (PCS) and
  Mental Component Summary (MCS).The higher the score, the worse the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, MD, Study Chair — Peking University People's Hospital
Locations (1):
- People's Hospital of Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No